CLINICAL TRIAL: NCT05078710
Title: A Pilot Study of Telitacicept Treatment in Primary APS Patients
Brief Title: Telitacicept in Primary APS Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: There is no clear therapeutic effect among the enrolled patients for the time being.
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-ZS-3026
Record Dates: First submitted 2021-09-24; First posted 2021-10-14 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2021-07

CONDITIONS: Anti Phospholipid Syndrome
Keywords: anti phospholipid syndrome
MeSH Terms: conditions — Antiphospholipid Syndrome | interventions — telitacicept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telitacicept arm (Experimental): Telitacicept 160mg once a week for 24 week as an add-on treatment regimen.
  Interventions: Drug: Telitacicept

INTERVENTIONS:
Drug: Telitacicept — 160mg once a week for 24 weeks
  Other Names: traditional antithrombotic and immunosuppressive treatment

SUMMARY:
This is a single-arm pilot study in Peking Union Medical College Hospital. Telitacicept will be added on traditional antithrombotic and immunosuppressive treatment in primary antiphospholipid syndrome (APS) patients with three positive antiphospholipid antibodies (aPL) and at least one extra-criteria manifestations, including thrombocytopenia, autoimmune hemolytic anemia, aPL associated nephropathy, heart valvular disease, non-stroke neurological manifestations. This study aims to evaluate the efficacy of Telitacicept in preventing thrombosis and improving extra-criteria manifestations on high-risk APS patients.

DETAILED DESCRIPTION:
The study started on July 2021 and will last 1.5 years. Primary APS patients with three positive aPL and extra-criteria manifestations with be enrolled. This is a single-arm pilot study. Telitacicept 160mg once a week for 24 weeks will be added on traditional antithrombotic and immunosuppressive treatment. Patients will be followed on week 12 and week 24. The primary endpoint is new thrombotic event. The secondary endpoints are improvement of extra-criteria manifestations, and titer change of aPL.

ELIGIBILITY:
Inclusion Criteria:

* meet 2006 Sapporo classification criteria of APS;
* diagnosis of primary APS, exclude other etiologies of thrombosis;
* with three aPL medium-to-high titer positivity, namely lupus anticoagulant, anti cardiolipin antibody, and anti-β2 glycoprotein antibody;
* with at least one extra-criteria manifestations of APS, including thrombocytopenia, hemolytic anemia, aPL nephropathy, valve heart disease and neurological manifestations.

Exclusion Criteria:

* overlap with other connective tissue diseases, such as systemic lupus erythematosus;
* during pregnancy;
* can not follow-up.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
new thrombotic event | 24 weeks
  any new thrombotic event during Telitacicept treatment

SECONDARY OUTCOMES:
improvement of thrombocytopenia during Telitacicept treatment | 24 weeks
  elevated platelet counts
improvement of hemolytic anemia during Telitacicept treatment | 24 weeks
  elevated hemoglobin
improvement of aPL nephropathy during Telitacicept treatment | 24 weeks
  decrease of proteinuria or creatinine
improvement of valve heart disease during Telitacicept treatment | 24 weeks
  decrease of valve thickness or vegetation by echocardiogram
improvement of neurological manifestations during Telitacicept treatment | 24 weeks
  MRI improvement
decrease of aPL titer during Telitacicept treatment | 24 weeks
  titer change of lupus anticoagulant, anticardiolipin antibody and anti-β2 glycoprotein-I antibody

CONTACTS AND LOCATIONS:
Overall Officials: Jiuliang Zhao, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No